CLINICAL TRIAL: NCT02437227
Title: A Phase 1, First in Man, Dual Centre, Open-label Dose Escalation Study With Expansion to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CCT3833 (BAL3833), a panRAF Inhibitor, Given Orally in Patients With Advanced Solid Tumours, Including Metastatic Melanoma
Brief Title: A Phase I, First in Man Study to Evaluate the Safety and Tolerability of a panRAF Inhibitor (CCT3833/BAL3833)in Patients With Solid Tumours
Acronym: PanRAF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other); Wellcome Trust (Other); Biomedical Research Centre for Cancer (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4232
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Melanoma; Cancer
MeSH Terms: conditions — Melanoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental: CCT3833 (Experimental): The starting dose of CCT3833 is 20 mg, taken as two 10 mg capsules. The starting schedule is a once daily continuous dosing schedule, but other dosing regimens may be considered depending on tolerability and exposures.The first dose of continuous dosing defines Cycle 1 Day 1. All treatment cycles have a duration of 28 days.
  Interventions: Drug: CCT3833

INTERVENTIONS:
Drug: CCT3833 — CCT3833 is a poorly soluble crystalline compound. It is multi-polymorphic and one form, designated Form D, has been purified and typically has a particle size of about 15-20 μm. Form D readily absorbs and desorbs water, but is not a hydrate and has been selected as the form to take forward into clinical development.

SUMMARY:
The study is a first in man, dose escalation study to evaluate the safety, tolerability and how the drug works in the body in patients with all solid tumours. The aim of this study is to determine the most effective dose of the study drug that can then be further investigated in patients with advanced melanoma.

DETAILED DESCRIPTION:
Metastatic malignant melanoma is the 5th most common cancer in the UK, with a notable proportion of young patients. The development of immunotherapies (such as Ipilimumab), and targeted therapies (such as Vemurafenib, a BRAF inhibitor) have resulted in improved survival outcomes for patients but is still only measured in months and not years. These targeted therapies are also only useful for patients with the relevant genetic mutation, leaving a significant proportion of patients without targeted therapy options. The need for more effective (and ideally curative) melanoma treatments remains. The Institute of Cancer Research, with funding from the Wellcome Trust, have created and developed a new panel of inhibitors that aim to more effectively terminate the growth, spread and survival signals that sustain the cancer. The broader targets allow patients possessing a range of genetic mutations to potentially benefit from this targeted therapy. It is hoped that these drugs could be used as both primary therapy for treatmentnaive patients as well as rescue therapy for those who have progressed on other targeted therapies.

This is a phase 1 study to evaluate the safety and effectiveness of one of these new compounds, CCT 3833, and to define the maximum tolerated dose in patients with advanced melanoma. The study also aims to examine the way that CCT3833 works within the body. Once the maximum tolerated dose has been established a small number of melanoma patients, with specific mutations and at different treatment option stages, will be treated to gain additional safety information and an initial indication of the possible efficacy of CCT3833 on melanoma tumours.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or over.
2. Written (signed and dated) informed consent and willing and capable of co-operating with study procedures, treatment and follow-up.
3. Histologically proven advanced or metastatic solid tumours.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Life expectancy of at least 12 weeks.
6. Haematological and biochemical indices (within 7 days before the first dose of CCT3833) within the ranges shown below:

   1. Haemoglobin (Hb) ≥ 9.0 g/dL.
   2. Absolute neutrophil count ≥ 1.5 x 109/L.
   3. Platelet count ≥ 100 x 109/L.
   4. Total bilirubin ≤ 1.5 x upper limit of normal (ULN), and Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x (ULN) (or ≤ 5 x ULN if elevated due to tumour).
   5. Calculated creatinine clearance > 50 mL/min (based on Cockcroft-Gault calculation).
7. Negative pregnancy test for females of child-bearing age.

Inclusion criteria: dose expansion cohort

Patients must meet ALL of the above criteria and additionally meet the following criteria:

1. Histologically proven locally advanced (unresectable) or metastatic melanoma.
2. Documented presence of either BRAF or RAS mutations, as established by validated mutation testing from tumour biopsy.
3. Evidence of measurable disease (according to RECIST v1.1)

Exclusion Criteria:

Patients who meet ANY of the following criteria will not be eligible to participate.

Patients who have had any of the following within the last 4 weeks:

1. Radiotherapy (except for palliative reasons), endocrine therapy (except luteinizing hormone releasing hormone (LHRH) agonists for prostate cancer), immunotherapy or chemotherapy (6 weeks for nitrosoureas, Mitomycin-C and 4 weeks for other investigational medicinal products (IMP)) before treatment. (For patients recruited to Part B (dose expansion) from Part A (dose escalation), prior treatment with CCT3833 during Part A (dose escalation) is permissible.)
2. Major surgery within the last four weeks.
3. Has been a participant in another interventional research study (involving an IMP) within the last 4 weeks, or plans to participate in one whilst taking part in this study. Participation in an observational study would be acceptable.

   Patients who have any of the following:
4. High medical risk because of non-malignant systemic disease including active, uncontrolled infection.
5. Known allergy to any pharmaceutical excipients.
6. Known to be serologically positive for Hepatitis B, Hepatitis C or Human Immunodeficiency Virus (HIV). Testing for these viruses is not mandatory.
7. Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

   1. History or presence of ventricular tachyarrhythmia.
   2. Presence of unstable atrial fibrillation (ventricular response > 100 bpm); patients with stable atrial fibrillation are eligible, provided they do not meet any of the other cardiac exclusion criteria.
   3. Repeated presence of a prolonged QTc interval > 450 ms at baseline (as calculated by Fridericia method).
   4. Unstable angina pectoris or acute myocardial infarction in the last 12 months prior to starting study drug.
   5. Other clinically significant heart disease (e.g., symptomatic congestive heart failure (LVEF < 50%); uncontrolled arrhythmia; history of labile hypertension or poor compliance with an antihypertensive regimen).
8. Uncontrolled hypertension that remains uncontrolled on > 1 antihypertensive agent.
9. Symptomatic brain metastases (if present they must have been stable for > 3 months). Such patients must not be requiring systemic corticosteroid or enzyme-inducing anticonvulsant therapy.
10. Inability to take oral medication; impairment of GI function or GI disease that could interfere with drug absorption.
11. Have taken potent inducers/inhibitors of CYP3A4 and CYP2C8 liver enzymes within 2 weeks of the first administration of study drug, or have conditions that require the concomitant usage of such drugs during the course of the study.
12. Are taking warfarin as an oral anticoagulant; patients anticoagulated with low molecular weight heparin are not excluded from the trial.
13. Female patients who are pregnant or lactating, or have the ability to become pregnant. However, those female patients who have a negative serum or urine pregnancy test before enrolment and are using highly-effective contraception during the study and for 6 months afterwards, are considered eligible. Highly-effective contraception methods include:

    1. Total abstinence.
    2. Male or female sterilization.
    3. A combination of any two of the following:

    i. Oral, injected or implanted hormonal contraception. ii. Placement of an intrauterine device (IUD) or intrauterine system (IUS). iii. Barrier methods of contraception: condom or diaphragm with spermicidal foam/gel/film/cream/vaginal suppository.
14. Male patients with partners of child-bearing potential, unless they agree to take measures not to father children by using one form of highly effective contraception as defined above, during the study and for 6 months afterwards. Men with pregnant or lactating partners should be advised to use barrier method contraception to prevent exposure to the foetus or neonate.
15. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Establishing the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of CCT3833. | 18 months
  The maximum tolerated dose is the dose at which no more than one patient out of up to six patients at the same dose level experience a highly probably or probably drug-related DLT as defined in the protocol. This dose level will be selected as the RP2D.
Assessing the safety and tolerability profile of CCT3833. (adverse event) | 18 months
  Determining causality of each adverse event (AE) to CCT3833 and grade according to NCI CTCAE v4.03.

SECONDARY OUTCOMES:
To determine the pharmacokinetic profile of CCT3833 in humans. (plasma levels of CCT3833) | 18 months
  Assessment of plasma levels of CCT3833 for 48 hours between Days -7 to -3 before Cycle 1, and on Cycle 2, Day 1.
To explore possible anti-tumour activity of CCT3833 in patients with advanced solid tumours.(measurable response (clinical or radiological) in any of the patients, as determined by the RECIST criteria v1.1) | 18 months
  Any measurable response (clinical or radiological) in any of the patients, as determined by the RECIST criteria v1.1.
Determining the correlation between PK exposures and tolerability and/or efficacy (i.e. defining the safe therapeutic range). | 18 months
  Correlation of plasma levels of CCT3833 with markers of efficacy and adverse event reports.

OTHER OUTCOMES:
To investigate the pharmacodynamic profile of CCT3833 in humans and to establish a biologically-active dose range. | 18 months
  Correlation of plasma levels of CCT3833 against tumour shrinkage data from imaging.
Determining magnitude and duration of effect in biomarkers (such as ERK, phosphorylated-ERK, Cyclin D1 and Ki-67) in surrogate and tumour tissue following CCT3833 administration. | 18 months
  Evaluation of a range of biomarkers from biopsies and optional blood biomarkers taken at baseline, on-treatment, and at disease progression.
Obtaining plasma samples for potential metabolite characterisation. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: James Larkin, Dr, Principal Investigator — Royla Marsden NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Christie NHS Foundation Trust, Manchester, Greater Manchester
  - Royal Marsden NHS Foundation Trust, Sutton, Surrey